CLINICAL TRIAL: NCT01146756
Title: Phase I Trial of the MEK Inhibitor AZD6244 in Combination With Thoracic Radiotherapy in Non-small Cell Lung Cancer
Brief Title: MEK Inhibitor and Thoracic Radiotherapy Trial
Acronym: MEKRT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Christie NHS Foundation Trust (Other)
Collaborators: AstraZeneca (Industry); University of Manchester (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09_DOG07_104
Record Dates: First submitted 2010-06-17; First posted 2010-06-22 (Estimated); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Non Small Cell Lung Cancer
Keywords: MEK inhibitor; thoracic radiotherapy; lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — AZD 6244

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AZD6244 & Thoracic Radiotherapy (Experimental): AZD6244 in combination with thoracic radiotherapy (RT)- the aim is to determine the recommended phase II dose (RP2D).
  Interventions: Drug: AZD6244

INTERVENTIONS:
Drug: AZD6244 — MEK inhibitor AZD6244 (Selumentinib) in combination with thoracic radiotherapy
  Other Names: Selumetinib

SUMMARY:
Two thirds of non small cell lung cancer patients present with locally advanced tumours (stage III) or metastatic disease (stage IV) and radiotherapy plays a major role in their treatment. Treatment (radiotherapy and chemotherapy) can be given with curative intent to selected patients with locally advanced, stage III disease. Patients with stage III tumours associated with a pleural effusion, and patients who present with advanced, metastatic disease (stage IV) are treated palliatively with no prospect of cure. In the latter, radiotherapy (RT) is offered with the aim of improving symptoms, achieving tumour control and optimising quality of life. It is generally believed that a plateau has been reached for combination of chemotherapy with radiotherapy lung cancer. There is a strong rationale for combining molecular targeted agents with irradiation. AZD6244 is a potent, selective, uncompetitive inhibitor of MEK that has been tested in early phase clinical trials either alone or in combination with chemotherapy in a variety of cancers including lung cancer. Preclinical studies have shown that AZD6244 enhances the effect of radiation. AZD6244 has not yet been combined with radiotherapy in clinical trials. In this study, a maximum of 18 patients will be allocated to one of 3 doses of AZD6244 in combination with a standard dose of RT in a Phase 1 dose escalation/ de-escalation design to determine the recommended dose for Phase 2 trials (RP2D). An expanded cohort of 15 patients will be treated at the RP2D to obtain additional safety and preliminary response data. Patients will undergo 3 FLT positron emission tomogram (PET) scans, the first scan before treatment, second scan during AZD6244 treatment and third scan during RT. All patients will also have tissue/blood samples collected for biomarkers. Biomarkers and FLTPET imaging will be examined to obtain information that may predict for response, resistance or toxicity to radiation and AZD6244.

DETAILED DESCRIPTION:
As above

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed NSCLC either inoperable, stage III NSCLC or stage IV NSCLC with dominant chest symptoms.
* Patient age ≥18
* Willingness and able to comply with treatment, tests and attend the required follow-up
* Prior chemotherapy is permitted provided the interval between day 8 of the last cycle of chemotherapy and day 1 of AZD6244 dosing is ≥2 weeks
* No prior radiotherapy or investigational agents
* Life expectancy estimated to be greater than 3 months
* Performance status(ECOG) 0 or 1
* MRC dyspnoea score <3
* Patient considered able to tolerate radical radiotherapy
* FEV1 >40% of predicted and DLCO (transfer factor for carbon monoxide) >40% of predicted
* Disease which can be encompassed within a radical radiotherapy treatment volume(V20 ≤35% and maximum cord dose 48Gy) on the radiotherapy planning scan
* Left ventricular ejection fraction >50% on baseline echocardiogram
* Adequate renal function - defined by GFR >50 ml/min (calculated Cockcroft and Gault) or by isotope GFR.
* Adequate bone marrow reserve: white cell count >3 x 109/l, absolute neutrophil count >1.5 x 109/l, haemoglobin >10.0 g/dl and platelet count >100 x 109/l (Blood transfusion permitted to achieve Hb >10g/dl)
* AST/ALT < 2.5 ULN and bilirubin <1.5 ULN
* Group D (expanded cohort) only: diameter of the primary tumour should be > 2 cm

Exclusion Criteria:

* Mixed non-small cell and small cell tumours
* Other previous or current malignant disease likely to interfere with protocol treatment or comparisons
* Lack of recovery from prior chemotherapy toxicity to grade ≤2 except alopecia d)Refractory nausea and vomiting, chronic gastrointestinal diseases (eg, inflammatory bowel disease), or significant bowel resection that would preclude adequate absorption of AZD6244
* Presence of clinically significant fluid accumulations in third spaces which cannot be adequately controlled by drainage or other procedures prior to inclusion in the study.
* History / evidence of active bleeding diatheses
* History of unstable diabetes
* History of interstitial pneumonitis
* Arterial hypertension defined as SBP≥ 160 or DBP ≥100 (antihypertensive medication to achieve these parameters are permissible)
* Myocardial infarction, or unstable or uncontrolled angina, congestive heart failure (NYHA > class II) within 1 year of enrollment
* Active infection on day of enrollment
* Uncontrolled hypercalcemia >3.0 or symptomatic
* History of hypersensitivity to active or inactive excipients of AZD6244
* Recent major surgery within 4 weeks prior to entry into the study (excluding the placement of vascular access) which would prevent administration of study treatment
* Known and symptomatic brain metastases. Brain imaging is not mandatory if patient is asymptomatic.
* Clinical judgement by the investigator that the patient should not participate in the study
* Patients of reproductive potential who are unable to comply with effective contraception if sexually active during the study and for a period of at least 90 days (men) or 6 months after treatment (women)
* Women who are breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2010-06-04 (Actual); Primary Completion 2017-02-08 (Actual); Study Completion 2017-02-08 (Actual)

PRIMARY OUTCOMES:
To determine the recommended phase II dose (RP2D) of AZD6244 in combination with thoracic radiotherapy (RT) | 18 months
  Recommended Phase II Dose (RP2D) - The RP2D will be the dose level at which < 2/6 patients experience dose limiting toxicity (DLT) during thoracic radiotherapy and for 12 weeks after completion of thoracic radiotherapy during the dose escalation phase. The RP2D will be further evaluated for safety in the expanded cohort.

SECONDARY OUTCOMES:
Secondary objectives : Safety profile of AZD6244 in combination with thoracic RT Dose delivery of AZD6244 in combination with thoracic RT Response to AZD6244 in combination with thoracic RT | 12 months
  Safety profile of AZD6244 in combination with thoracic RT. Dose delivery of AZD6244 in combination with thoracic RT. Response to AZD6244 in combination with thoracic RT

CONTACTS AND LOCATIONS:
Overall Officials: Corinne Faivre-Finn, MD, PhD, Principal Investigator — The Christie NHS Foundation Trust
Locations (1):
- The Christie NHS Foundation Trust, Manchester, Greater Manchester, United Kingdom

REFERENCES:
- [Derived] Haslett K, Koh P, Hudson A, Ryder WD, Falk S, Mullan D, Taylor B, Califano R, Blackhall F, Faivre-Finn C. Phase I trial of the MEK inhibitor selumetinib in combination with thoracic radiotherapy in non-small cell lung cancer. Clin Transl Radiat Oncol. 2021 Feb 25;28:24-31. doi: 10.1016/j.ctro.2021.02.008. eCollection 2021 May. PMID 33748440
- See also: One of Europe's leading cancer centres — http://www.christie.nhs.uk